CLINICAL TRIAL: NCT01309217
Title: Dissemination of Tobacco Tactics Versus 1-800-QUIT-NOW for Hospitalized Smokers
Brief Title: Dissemination of Tobacco Tactics for Hospitalized Smokers
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Sonia Duffy, Associate Professor, University of Michigan
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 1U01HL105218-01 (NIH)
Record Dates: First submitted 2011-03-04; First posted 2011-03-07 (Estimated); Last update posted 2014-11-18 (Estimated); Status verified 2014-11

CONDITIONS: Smoking Cessation
MeSH Terms: conditions — Smoking Cessation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Usual Care (Active Comparator): The comparison group will receive usual care in accordance to how the hospital responds to current Joint Commission on Accreditation of Healthcare Organization's (JC) standards. See below for a complete description.
  Interventions: Other: Usual Care
- Tobacco Tactics Intervention (Experimental): At the intervention sites the research nurse will teach the Tobacco Tactics Intervention to nurses. For nurses, the Cessation Toolkit includes: 1) 1 CEU contact hour for training; 2) PowerPoint presentation on behavioral and pharmaceutical interventions; 3) pocket card "Helping Smokers Quit: A Guide for Clinicians" developed by U.S. Department of Health and Human Services, Public Health Service; 4) behavioral and pharmaceutical protocols; and 5) computerized template for nurse documentation. For patients, the Cessation Toolkit includes: 1) brochure; 2) videotape; 3); and 4) pharmaceuticals.
  Interventions: Behavioral: Tobacco Tactics Intervention

INTERVENTIONS:
Behavioral: Tobacco Tactics Intervention — At the intervention sites the research nurse will teach the Tobacco Tactics Intervention to nurses. For nurses, the Cessation Toolkit includes: 1) 1 CEU contact hour for training; 2) PowerPoint presentation on behavioral and pharmaceutical interventions; 3) pocket card "Helping Smokers Quit: A Guide for Clinicians" developed by U.S. Department of Health and Human Services, Public Health Service; 4) behavioral and pharmaceutical protocols; and 5) computerized template for nurse documentation. For patients, the Cessation Toolkit includes: 1) brochure; 2) videotape; 3); and 4) pharmaceuticals.
  Arms: Tobacco Tactics Intervention
Other: Usual Care — The comparison group will receive usual care in accordance to how the hospital responds to current Joint Commission on Accreditation of Healthcare Organization's (JC) standards. JC standards require that a patient with a smoking history receives at least one of the following: advice to stop smoking, brochures or handouts on smoking cessation, a smoking cessation aid such as nicotine patch, gum, nasal spray, inhaler, lozenge, or bupropion SR, viewed a smoking cessation video.
  Arms: Usual Care

SUMMARY:
Nurse-administered smoking cessation interventions have been shown to be efficacious, but are seldom implemented due to lack of training and time. This project aims to disseminate and test the nurse-administered Tobacco Tactics intervention in 6 hospitals.

DETAILED DESCRIPTION:
Background: Dr. Duffy has developed, tested, and refined the efficacious, nurse-administered Tobacco Tactics intervention and has packaged it into a Toolkit for dissemination in two Veterans Affairs (VA) hospitals. However, rigorous testing of dissemination outside of the VA is needed.

Objectives: Using 6 community hospitals in the Trinity Health System, the objectives of this study are to:

1. Determine provider and patient receptivity, barriers, and facilitators to implementing the nurse-administered, inpatient Tobacco Tactics intervention versus usual care using face-to-face feedback and surveys.
2. Compare the effectiveness of the nurse-administered, inpatient Tobacco Tactics intervention versus usual care across hospitals, units, and patient characteristics using biochemically confirmed 7-day point-prevalence abstinence at 6-month cessation as the primary outcome.
3. Determine the cost-effectiveness of the nurse-administered, inpatient Tobacco Tactics intervention versus usual care including the cost per quitter, cost per life-year saved, and cost per quality-adjusted life-year saved.

Methods: This effectiveness study will be a cluster randomized control trial in 6 Michigan community hospitals of which 3 will get the nurse-administered Tobacco Tactics intervention and the other 3 will provide their usual care in accordance to how the hospital responds to current Joint Commission on Accreditation of Healthcare Organization's (JC) standards. A research nurse will disseminate the intervention in the 3 out of 6 sites to Master Trainers who will teach staff nurses on all shifts on all units, until all staff nurses are trained. The interventions will become the standard of care within the intervention sites. Research nurses will also conduct rolling evaluation to identify barriers and facilitators to dissemination and implement measures to ensure sustainability of the intervention. It is expected that 7,868 inpatient smokers per year will be eligible to participate in the study of which the investigators expect to recruit 2,350 to have sufficient power to analyze the objectives. Descriptive statistics (means and frequency distributions) will be used to summarize the nurses' survey results, participation rates, smokers' receipt of specific cessation services, and satisfaction with services. Logistic regressions and t-tests will be used to determine differences between intervention groups on satisfaction and quit rates, respectively, with adjustment for the clustering of patients within units and hospitals. Regression analyses will test the moderation of the effects of the interventions by patient characteristics such as confidence in ability to quit, nicotine addiction, alcohol intake, depression, demographics and a smoking related diagnosis such as heart disease. Cost-effectiveness will be assessed by constructing 3 ratios including the cost per quitter, cost per life-year saved, and the cost per quality-adjusted life-year saved.

ELIGIBILITY:
Inclusion Criteria:

1. are at least 18 years of age;
2. have smoked within one month prior to hospitalization;
3. have a projected hospital stay of at least 24 hours; and
4. are willing to complete the interview surveys.

Exclusion Criteria:

1. are too ill to participate;
2. are terminal;
3. are involved in a concurrent trial that includes intervention on smoking; and
4. are non-English speaking (the intervention is currently only in English);
5. have significant cognitive impairment; and
6. have significant communication barriers.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1528 (Actual)
Dates: Start 2011-07; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Biochemically confirmed 7-day point-prevalence abstinence at 6-month | 6-month follow-up
  The question used to evaluate smoking is: "Have you smoked any cigarette products, even a puff, in the last seven days?" Along with the 6-month survey, patients will be sent a sample for NicAlert urinary test.

CONTACTS AND LOCATIONS:
Overall Officials: Sonia A Duffy, PhD, RN, Principal Investigator — University of Michigan
Locations (6):
- United States (6):
  - Saint Mary's Healthcare, Grand Rapids, Michigan
  - St. Mary Mercy, Livonia, Michigan
  - Mercy Health Partners - Hackley Campus, Muskegon, Michigan
  - Mercy Health Partners - Mercy Campus, Muskegon, Michigan
  - St. Joseph Mercy, Oakland, Michigan
  - St. Joseph Mercy Hospital, Ypsilanti, Michigan

REFERENCES:
- [Background] Duffy SA, Reeves P, Hermann C, Karvonen C, Smith P. In-hospital smoking cessation programs: what do VA patients and staff want and need? Appl Nurs Res. 2008 Nov;21(4):199-206. doi: 10.1016/j.apnr.2006.11.002. PMID 18995161
- [Background] Freund M, Campbell E, Paul C, McElduff P, Walsh RA, Sakrouge R, Wiggers J, Knight J. Smoking care provision in hospitals: a review of prevalence. Nicotine Tob Res. 2008 May;10(5):757-74. doi: 10.1080/14622200802027131. PMID 18569750
- [Background] Rice VH, Stead LF. Nursing interventions for smoking cessation. Cochrane Database Syst Rev. 2004;(1):CD001188. doi: 10.1002/14651858.CD001188.pub2. PMID 14973964
- [Background] Duffy SA, Ronis DL, Valenstein M, Lambert MT, Fowler KE, Gregory L, Bishop C, Myers LL, Blow FC, Terrell JE. A tailored smoking, alcohol, and depression intervention for head and neck cancer patients. Cancer Epidemiol Biomarkers Prev. 2006 Nov;15(11):2203-8. doi: 10.1158/1055-9965.EPI-05-0880. PMID 17119047
- [Background] Duffy SA, Karvonen-Gutierrez CA, Ewing LA, Smith PM; Veterans Integrated Services Network 11 Tobacco Tactics Team. Implementation of the Tobacco Tactics program in the Department of Veterans Affairs. J Gen Intern Med. 2010 Jan;25 Suppl 1(Suppl 1):3-10. doi: 10.1007/s11606-009-1075-9. PMID 20077145
- [Background] Rigotti NA, Munafo MR, Stead LF. Smoking cessation interventions for hospitalized smokers: a systematic review. Arch Intern Med. 2008 Oct 13;168(18):1950-60. doi: 10.1001/archinte.168.18.1950. PMID 18852395
- [Background] Rice VH, Stead LF. Nursing interventions for smoking cessation. Cochrane Database Syst Rev. 2008 Jan 23;(1):CD001188. doi: 10.1002/14651858.CD001188.pub3. PMID 18253987
- [Background] Rice VH. Nursing intervention and smoking cessation: A meta-analysis. Heart Lung. 1999 Nov-Dec;28(6):438-54. doi: 10.1016/s0147-9563(99)70033-6. PMID 10580218
- [Background] Terrell JE, Ronis DL, Fowler KE, Bradford CR, Chepeha DB, Prince ME, Teknos TN, Wolf GT, Duffy SA. Clinical predictors of quality of life in patients with head and neck cancer. Arch Otolaryngol Head Neck Surg. 2004 Apr;130(4):401-8. doi: 10.1001/archotol.130.4.401. PMID 15096421
- [Background] Duffy SA, Ronis DL, Valenstein M, Fowler KE, Lambert MT, Bishop C, Terrell JE. Depressive symptoms, smoking, drinking, and quality of life among head and neck cancer patients. Psychosomatics. 2007 Mar-Apr;48(2):142-8. doi: 10.1176/appi.psy.48.2.142. PMID 17329608
- [Background] Etter JF, Bergman MM, Humair JP, Perneger TV. Development and validation of a scale measuring self-efficacy of current and former smokers. Addiction. 2000 Jun;95(6):901-13. doi: 10.1046/j.1360-0443.2000.9569017.x. PMID 10946439
- [Background] Cohen S, Lichtenstein E. Partner behaviors that support quitting smoking. J Consult Clin Psychol. 1990 Jun;58(3):304-9. doi: 10.1037//0022-006x.58.3.304. PMID 2365893
- [Background] Cohen S, Kamarck T, Mermelstein R. A global measure of perceived stress. J Health Soc Behav. 1983 Dec;24(4):385-96. No abstract available. PMID 6668417
- [Background] Rigotti NA, Munafo MR, Stead LF. Interventions for smoking cessation in hospitalised patients. Cochrane Database Syst Rev. 2007 Jul 18;(3):CD001837. doi: 10.1002/14651858.CD001837.pub2. PMID 17636688
- [Background] Saunders JB, Aasland OG, Babor TF, de la Fuente JR, Grant M. Development of the Alcohol Use Disorders Identification Test (AUDIT): WHO Collaborative Project on Early Detection of Persons with Harmful Alcohol Consumption--II. Addiction. 1993 Jun;88(6):791-804. doi: 10.1111/j.1360-0443.1993.tb02093.x. PMID 8329970
- [Background] Stump TE, Clark DO, Johnson RJ, Wolinsky FD. The structure of health status among Hispanic, African American, and white older adults. J Gerontol B Psychol Sci Soc Sci. 1997 May;52 Spec No:49-60. doi: 10.1093/geronb/52b.special_issue.49. PMID 9215357
- [Background] Simon JA, Solkowitz SN, Carmody TP, Browner WS. Smoking cessation after surgery. A randomized trial. Arch Intern Med. 1997 Jun 23;157(12):1371-6. PMID 9201012
- [Background] Chen Y, Rennie DC, Dosman JA. The reliability of cigarette consumption reports by spousal proxies. Am J Public Health. 1995 Dec;85(12):1711-2. doi: 10.2105/ajph.85.12.1711. No abstract available. PMID 7503354
- [Background] Fagerstrom KO, Heatherton TF, Kozlowski LT. Nicotine addiction and its assessment. Ear Nose Throat J. 1990 Nov;69(11):763-5. No abstract available. PMID 2276350
- [Background] Smith MW, Barnett PG. Direct measurement of health care costs. Med Care Res Rev. 2003 Sep;60(3 Suppl):74S-91S. doi: 10.1177/1077558703257001. PMID 15095547
- [Background] Golding JM, Gongla P, Brownell A. Feasibility of validating survey self-reports of mental health service use. Am J Community Psychol. 1988 Feb;16(1):39-51. doi: 10.1007/BF00906071. PMID 3369382
- [Background] Weissman JS, Levin K, Chasan-Taber S, Massagli MP, Seage GR 3rd, Scampini L. The validity of self-reported health-care utilization by AIDS patients. AIDS. 1996 Jun;10(7):775-83. doi: 10.1097/00002030-199606001-00013. PMID 8805870
- [Background] Thompson BT, Schoenfeld D. Usual care as the control group in clinical trials of nonpharmacologic interventions. Proc Am Thorac Soc. 2007 Oct 1;4(7):577-82. doi: 10.1513/pats.200706-072JK. PMID 17878473
- [Background] Lindquist R, Wyman JF, Talley KM, Findorff MJ, Gross CR. Design of control-group conditions in clinical trials of behavioral interventions. J Nurs Scholarsh. 2007;39(3):214-21. doi: 10.1111/j.1547-5069.2007.00171.x. PMID 17760793
- [Background] Kottke TE, Battista RN, DeFriese GH, Brekke ML. Attributes of successful smoking cessation interventions in medical practice. A meta-analysis of 39 controlled trials. JAMA. 1988 May 20;259(19):2883-9. doi: 10.1001/jama.259.19.2883. PMID 3367456
- [Background] Lancaster T, Stead L. Physician advice for smoking cessation. Cochrane Database Syst Rev. 2004 Oct 18;(4):CD000165. doi: 10.1002/14651858.CD000165.pub2. PMID 15494989
- [Background] An LC, Zhu SH, Nelson DB, Arikian NJ, Nugent S, Partin MR, Joseph AM. Benefits of telephone care over primary care for smoking cessation: a randomized trial. Arch Intern Med. 2006 Mar 13;166(5):536-42. doi: 10.1001/archinte.166.5.536. PMID 16534040
- [Background] Lichtenstein E, Glasgow RE, Lando HA, Ossip-Klein DJ, Boles SM. Telephone counseling for smoking cessation: rationales and meta-analytic review of evidence. Health Educ Res. 1996 Jun;11(2):243-57. doi: 10.1093/her/11.2.243. PMID 10163409
- [Background] Smith PM, Cameron R, McDonald PW, Kawash B, Madill C, Brown KS. Telephone counseling for population-based smoking cessation. Am J Health Behav. 2004 May-Jun;28(3):231-41. doi: 10.5993/ajhb.28.3.4. PMID 15152882
- [Background] Wilson W, Pratt C. The impact of diabetes education and peer support upon weight and glycemic control of elderly persons with noninsulin dependent diabetes mellitus (NIDDM). Am J Public Health. 1987 May;77(5):634-5. doi: 10.2105/ajph.77.5.634. PMID 3565666
- [Background] Thomson O'Brien MA, Freemantle N, Oxman AD, Wolf F, Davis DA, Herrin J. Continuing education meetings and workshops: effects on professional practice and health care outcomes. Cochrane Database Syst Rev. 2001;(2):CD003030. doi: 10.1002/14651858.CD003030. PMID 11406063
- [Background] McAlister AL, Rabius V, Geiger A, Glynn TJ, Huang P, Todd R. Telephone assistance for smoking cessation: one year cost effectiveness estimations. Tob Control. 2004 Mar;13(1):85-6. doi: 10.1136/tc.2003.004515. PMID 14985603
- [Background] Javitz HS, Swan GE, Zbikowski SM, Curry SJ, McAfee TA, Decker DL, Patterson R, Jack LM. Cost-effectiveness of different combinations of bupropion SR dose and behavioral treatment for smoking cessation: a societal perspective. Am J Manag Care. 2004 Mar;10(3):217-26. PMID 15032259
- [Derived] Duffy SA, Ronis DL, Ewing LA, Waltje AH, Hall SV, Thomas PL, Olree CM, Maguire KA, Friedman L, Klotz S, Jordan N, Landstrom GL. Implementation of the Tobacco Tactics intervention versus usual care in Trinity Health community hospitals. Implement Sci. 2016 Nov 4;11(1):147. doi: 10.1186/s13012-016-0511-6. PMID 27814722
- [Derived] Duffy SA, Ronis DL, Karvonen-Gutierrez CA, Ewing LA, Hall SV, Yang JJ, Thomas PL, Olree CM, Maguire KA, Friedman L, Gray D, Jordan N. Effectiveness of the Tobacco Tactics Program in the Trinity Health System. Am J Prev Med. 2016 Oct;51(4):551-65. doi: 10.1016/j.amepre.2016.03.012. PMID 27647056
- [Derived] Duffy SA, Cummins SE, Fellows JL, Harrington KF, Kirby C, Rogers E, Scheuermann TS, Tindle HA, Waltje AH; Consortium of Hospitals Advancing Research on Tobacco (CHART). Fidelity monitoring across the seven studies in the Consortium of Hospitals Advancing Research on Tobacco (CHART). Tob Induc Dis. 2015 Sep 3;13(1):29. doi: 10.1186/s12971-015-0056-5. eCollection 2015. PMID 26336372
- [Derived] Duffy SA, Ronis DL, Titler MG, Blow FC, Jordan N, Thomas PL, Landstrom GL, Ewing LA, Waltje AH. Dissemination of the nurse-administered Tobacco Tactics intervention versus usual care in six Trinity community hospitals: study protocol for a comparative effectiveness trial. Trials. 2012 Aug 1;13:125. doi: 10.1186/1745-6215-13-125. PMID 22852834